CLINICAL TRIAL: NCT04508465
Title: Persistent Postoperative Pain After Major Emergency Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Cecilie Bauer Derby, Research coordinator RN, Zealand University Hospital
Other Study IDs: 2020
Record Dates: First submitted 2020-07-30; First posted 2020-08-11 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OMEGA: Patients who have undergone major emergency abdominal surgery including the stomach, small or large bowel, or rectum for conditions such as perforation, ischemia, abdominal abscess, bleeding or obstruction.

SUMMARY:
Perioperative pain is one of the most significant complaints and problems for patients undergoing major open surgery. Pain after surgery carry an abundance of consequences such as reduced mobilization, reduced nutrition intake, reduced pulmonary capacity and increased risk of complications and length of hospitalization. The literature does not supply much information on short- or longer-term outcomes of pain treatment for emergency surgery. The investigators know that for planned surgery in general around 10-50 percentage suffer from persistent postoperative pain. It is therefore important to follow-up on the longer-term outcomes after the standardized analgesic pain treatment. Based on a predefined patient group called OMEGA (Optimizing Major EMergency Abdominal surgery) the investigators hypothesize that OMEGA patients will present a significant incidence rate of patients with persistent postoperative pain and/or continued opioid/non-opioid usage. Therefore this study is to investigate the incidence of prolonged postoperative pain and opioid/non-opioid consumption in OMEGA patients at 3 month after major emergency abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* OMEGA patients (patients who have undergone major emergency abdominal surgery including the stomach, small or large bowel, or rectum for conditions such as perforation, ischemia, abdominal abscess, bleeding or obstruction)
* Age 18 or more
* Surgery performed within 72 hours of an acute admission or as an acute re-operation

Exclusion Criteria:

* Elective laparoscopy
* Diagnostic laparotomy/laparoscopy where no subsequent procedure is performed
* Non-elective hernia repair without bowel resection
* Admission or transfer to an intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone major emergency abdominal surgery at the department of abdominal surgery at Zealand University Hospital Køge
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-03-04 (Estimated); Study Completion 2021-06-04 (Estimated)

PRIMARY OUTCOMES:
Pain Mobilization | Data is collected 3 months postoperative
  Pain during mobilization last week based on a self-made questionary
Opioids | Data is collected 3 months postoperative
  Daily opioid usage last week based on a self-made questionary

SECONDARY OUTCOMES:
Pain Rest | Data is collected 3 months postoperative
  Pain in rest last week based on a self-made questionary
Non-opiod Analgesic | Data is collected 3 months postoperative
  Non-opioid analgesic usage based on a self-made questionary
Barthel-20 Index | Data is collected 3 months postoperative
  Simple function measurement based on daily living
  Simple function measurement
EuroQol-5 | Data is collected 3 months postoperative
  Health related quality of life
Montreal Cognitive Assessment test (Mini-MoCA) | Data is collected 3 months postoperative
  Cognitive function

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Department of Anaesthesiology, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No